CLINICAL TRIAL: NCT05588167
Title: Establishment of Genomic and Phenotypic Database for Niemann-Pick Disease, Type C
Status: Recruiting | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001018; 001018-CH
Record Dates: First submitted 2022-10-19; First posted 2022-10-20 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-03-19

CONDITIONS: Niemann-Pick Disease, Type C
Keywords: Genetic; Clinical; DNA; Medical; History; Natural History
MeSH Terms: conditions — Niemann-Pick Disease, Type C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Affected: Patients with Niemann-Pick Disease, type C

SUMMARY:
Background:

Niemann-Pick type C (NPC) disease is a rare, progressive neurodegenerative disease that affects mainly the brain, liver, and spleen but also other parts of the body. There is no cure for NPC, and symptoms only get worse over time. Symptoms can include seizures, difficulty moving or talking, or dementia. But symptoms can vary among different people with the disease. Some may have seizures, while others do not, for example. Some people begin showing symptoms in childhood; in others, symptoms may not appear until they are adults. Researchers want to learn more about why NPC affects people differently. This natural history study will gather data from people with NPC in order to understand more about the disease and how it affects the body.

Objective:

This study will create the first and largest database about NPC.

Eligibility:

People of any age who have NPC.

Design:

Participants will have blood drawn from a vein. This will happen only once. The blood will be used to analyze the participants DNA.

The participants medical records will be reviewed. The study team will collect data on participants NPC diagnosis and symptoms; they will record how long participants have had each symptom. The study team will also collect data on each participants age, sex, race, height, weight, medications, and other test results.

The study team will communicate with participants. They will discuss the study and answer any questions.

Participants will receive up to $190.

...

DETAILED DESCRIPTION:
Study Description:

The primary objective of this protocol is to investigate the phenotypic heterogeneity of NPC by using clinical and genomic data, and to establish a comprehensive database to facilitate future investigations.

Objectives:

1. Identify correlations between NPC clinical phenotypic findings and genomic markers to facilitate the understanding of the heterogeneity of this disease.
2. Identify genetic contributions to NPC disease progression that can be utilized as potential therapeutic targets.
3. Establish the first and largest database of genomic and phenotypic information for NPC to benefit the NPC research and patient community.

ELIGIBILITY:
* INCLUSION CRITERIA;

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, any age, demographic or ethnic background will be eligible for this study
4. Diagnosis of NPC will be based on clinical, biochemical or molecular testing.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Unwilling to provide consent
2. Unable to provide biospecimen to obtain DNA
3. Unable to provide medical records or clinical data

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with Niemann-Pick Disease, type C
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical data, genomic markers | 2 years
  Identify correlations between NPC clinical phenotypic findings and genomic markers to facilitate the understanding of the heterogeneity of this disease.
Whole genome | 2 years
  Identify genetic contributions to NPC disease progression that can be utilized as potential therapeutic targets.

CONTACTS AND LOCATIONS:
Overall Officials: Forbes D Porter, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001018-CH.html